CLINICAL TRIAL: NCT06884423
Title: Infant Survival and Long-term Outcome Following Fetoscopic Endoluminal Tracheal Occlusion in Severe Left and Right Congenital Diaphragmatic Hernia, A Phase III Trial
Brief Title: Safety and Efficacy of FETO in CDH: A Phase III Trial
Acronym: CHOP FETO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Holly L Hedrick, MD (Other)
Responsible Party: Sponsor-Investigator, Holly L Hedrick, MD, Sponsor-Investigator, Attending Surgeon, Professor of Surgery, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-022603; G140236 (Other: U.S. Food and Drug Administration)
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Congenital Diaphragmatic Hernia; Pulmonary Hypoplasia
Keywords: congenital diaphragmatic hernia; tracheal occlusion
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- FETO in CDH (Experimental): Fetoscopic Endoluminal Tracheal Occlusion (FETO) will be performed by placing a detachable balloon inside the fetal airway and removing the balloon after several weeks. Devices: GoldBAL2 Detachable Balloon and BALTACCIBDPE100 Delivery Catheter. Assignment will be non-randomized. 40 maternal/fetal dyads will be enrolled in this arm.
  Interventions: Device: FETO with GoldBAL2 Balloon and BALTACCIBDPE100 Catheter
- Expectant Management in CDH (No Intervention): The control arm includes patients eligible for FETO according to side of defect, O/E LHR, and liver position who undergo expectant management rather than FETO intervention. Assignment will be non-randomized. 40 maternal/fetal dyads will be enrolled in this arm.

INTERVENTIONS:
Device: FETO with GoldBAL2 Balloon and BALTACCIBDPE100 Catheter — Fetoscopic Endoluminal Tracheal Occlusion (FETO) in CDH with GoldBAL2 Detachable Balloon and BALTACCIBDPE100 Delivery Catheter
  Arms: FETO in CDH

SUMMARY:
Congenital diaphragmatic hernia (CDH) is a birth defect characterized by the development of a hole in the diaphragm, the breathing muscle that separates the chest from the abdomen. As a result, organs in the abdomen can move into the chest and press on the developing lungs. This prevents the lungs from growing and developing normally.

In severe cases, CDH can lead to serious disease and death at birth. For these babies, treatment before birth may allow the lungs to grow enough before birth so these children are capable of surviving and thriving.

DETAILED DESCRIPTION:
All patients will complete a standard prenatal evaluation at the Children's Hospital of Philadelphia (CHOP) Center for Fetal Diagnosis and Treatment (CFDT) to determine if they are candidates for this study. The standard clinical assessments include medical history and physical exam, level II ultrasound, fetal echocardiogram, fetal magnetic resonance imaging (MRI), and a psychosocial assessment.

If determined eligible for fetoscopic endoluminal tracheal occlusion (FETO) intervention, patients will be extensively counseled by the CFDT Team and those who choose to participate will provide written, informed consent for study enrollment.

Up to 40 maternal/fetal dyads will be enrolled in the intervention arm of this study. The pregnant patient and fetus will undergo two procedures. A balloon will be placed in the fetal airway between 27+0/7 - 29+6/7 gestational age. The balloon blocks the airway and remains in place until balloon removal. The timing for balloon removal will be determined by the CFDT Management Team and can occur between 34 +0/7 - 34+6/7 gestational age.

Pregnant patients enrolled in the intervention arm of study must remain near the fetal center, under close supervision, from the time of balloon placement through delivery in the CHOP Garbose Family Special Delivery Unit.

Weekly prenatal monitoring will occur after the first procedure at the CFDT, and planned delivery will occur in the Garbose Family Special Delivery Unit at term.

Postnatal stabilization and subsequent surgery to repair the diaphragm will take place at CHOP.

Up to 40 maternal/fetal dyads which meet criteria according to defect side, observed/expected lung to head ratio (O/E LHR), and liver position, but undergo expectant management rather than FETO intervention, will be enrolled in the control arm of this study.

Infants in both the intervention arm and the control arm will be followed at CHOP at 6 months, 12 months, 18 months, and 24 months of age through the CHOP Pulmonary Hypoplasia Program.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women age 18 years and older
2. Singleton pregnancy
3. Normal fetal karyotype with confirmation by culture results, whole exome sequencing (WES), whole genome sequencing (WGS), or chromosomal microarray with non-pathologic variants. Results by fluorescence in situ hybridization (FISH) will be acceptable if the patient is greater than 26 weeks.
4. Gestational age at enrollment is prior to 29 weeks 6 days
5. Liver is intrathoracic
6. Isolated left congenital diaphragmatic hernia (CDH) with observed/expected lung to head ratio (O/E LHR) of less than 30% at enrollment (18^0 to 29^5 weeks), or:
7. Isolated right CDH with O/E LHR equal to or less than 45% at enrollment (18^0 to 29^5 weeks).
8. Cervical length by transvaginal ultrasound equal to or greater than 20 mm within 24 hours of fetoscopic endoluminal tracheal occlusion (FETO) procedure
9. Patient meets psychosocial criteria
10. Informed consent

Exclusion Criteria:

1. Patient is less than 18 years of age
2. Multi-fetal pregnancy
3. History of natural rubber latex allergy
4. Preterm labor, cervix shortened (less than 20 mm at enrollment or within 24 hours of FETO balloon insertion procedure) or uterine anomaly strongly predisposing to preterm labor, placenta previa
5. Psychosocial ineligibility, precluding consent:

   * Inability to reside within 30 minutes of the Children's Hospital of Philadelphia (CHOP) and inability to comply with the travel for the follow-up requirements of the trial
   * Patient does not have a support person (e.g. spouse, partner, mother) available to stay with the patient for the duration of the pregnancy at CHOP
6. Bilateral CDH, isolated left sided CDH with O/E LHR greater than or equal to 30% (measured at 18^0 to 29^5 weeks), isolated right sided CDH with O/E LHR greater than 45% (measured at 180 to 295 weeks), as determined by ultrasound
7. No Liver herniation into thoracic cavity.
8. Additional fetal anomaly by ultrasound, magnetic resonance imaging (MRI), or echocardiogram at the fetal treatment center. Exclude chromosomal abnormalities, associated anomalies recognized to alter survival prognosis (ie. CDH and congenital heart disease) or presence of an underlying genetic syndrome (ie. Fryns).
9. Maternal contraindication to fetoscopic surgery or severe maternal medical condition in pregnancy
10. History of incompetent cervix with or without cerclage
11. Placental abnormalities (previa, abruption, accrete) known at time of enrollment.
12. Maternal-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy.
13. Maternal HIV, Hepatitis-B, Hepatitis-C status positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patient's HIV or Hepatitis status is unknown, the patient must be tested and found to have negative results before enrollment.
14. Uterine anomaly such as large or multiple fibroids or mullerian duct abnormality
15. There is no safe or technically feasible fetoscopic approach to balloon placement.
16. Participation in another intervention study that influences maternal and fetal morbidity and mortality or participation in this trial in a previous pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Successful placement and removal of the FETO Device | 24 months
  Evalutation of successful placement and removal of the fetoscopic endoluminal tracheal occlusion (FETO) device in cases of intrathoracic liver herniation with isolated left congenital diaphragmatic hernia (LCDH) with observed/expected lung to head ratio (O/E LHR) < 30% or isolated right congenital diaphragmatic hernia (RCDH) with O/E LHR < 45%.
Comparison of neonatal survival rates of LCDH cases between intervention and control groups | 24 months
  Compare survival to discharge from the neonatal intensive care units (NICU), between fetuses with intrathoracic liver herniation and isolated LCDH with O/E LHR < 30% that receive FETO procedure performed at 27^0 to 29^6 weeks gestation to concurrent patients with intrathoracic liver herniation, isolated LCDH and O/E LRH < 30% that undergo expectant management.
Comparison of neonatal survival rates of RCDH cases between intervention and control groups | 24 months
  Compare the neonatal survival rate to discharge from the neonatal intensive care units (NICU), between fetuses with intrathoracic liver herniation, isolated RCDH with O/E LHR < 45% that undergo FETO procedure performed at 27^0 to 29^6 weeks gestation to concurrent patients with intrathoracic liver herniation, isolated RCDH and O/E LHR < 45% that proceed with expectant management.
Assessment of complications associated with the FETO intervention | 24 months
  Evaluate the frequency of maternal and fetal complications associated with the FETO intervention.

SECONDARY OUTCOMES:
Comparison of long-term mortality and morbidity of LCDH cases between intervention and control groups | 24 months
  Evaluate whether the FETO procedure is associated with reduced long-term mortality and morbidities at 6, 12, 18 and 24 months in isolated LCDH survivors with O/E LHR < 30% when compared to concurrent isolated LCDH with O/E LRH < 30% that undergo expectant management where all fetuses were found to have intrathoracic liver herniation.
Comparison of long-term mortality and morbidity of RCDH cases between intervention and control groups | 24 months
  Evaluate whether the FETO procedure is associated with reduced long-term mortality and morbidities at 6, 12, 18, and 24 months in isolated RCDH survivors with O/E LHR ≤ 45% when compared to concurrent isolated RCDH with LHR ≤ 45% that undergo expectant management where all fetuses were found to have intrathoracic liver herniation.

CONTACTS AND LOCATIONS:
Overall Officials: Holly L Hedrick, MD, FACS, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A deidentified data set will be shared with other NAFTNet institutions which perform FETO. These data will be shared under a data sharing agreement.

REFERENCES:
- [Background] Danzer E, Hedrick HL. Controversies in the management of severe congenital diaphragmatic hernia. Semin Fetal Neonatal Med. 2014 Dec;19(6):376-84. doi: 10.1016/j.siny.2014.10.001. Epub 2014 Nov 7. PMID 25454678
- [Background] Deprest JA, Gratacos E, Nicolaides K, Done E, Van Mieghem T, Gucciardo L, Claus F, Debeer A, Allegaert K, Reiss I, Tibboel D. Changing perspectives on the perinatal management of isolated congenital diaphragmatic hernia in Europe. Clin Perinatol. 2009 Jun;36(2):329-47, ix. doi: 10.1016/j.clp.2009.03.004. PMID 19559323
- [Background] Jani JC, Nicolaides KH, Gratacos E, Valencia CM, Done E, Martinez JM, Gucciardo L, Cruz R, Deprest JA. Severe diaphragmatic hernia treated by fetal endoscopic tracheal occlusion. Ultrasound Obstet Gynecol. 2009 Sep;34(3):304-10. doi: 10.1002/uog.6450. PMID 19658113
- [Background] Style CC, Olutoye OO, Belfort MA, Ayres NA, Cruz SM, Lau PE, Shamshirsaz AA, Lee TC, Olutoye OA, Fernandes CJ, Cortes MS, Keswani SG, Espinoza J. Fetal endoscopic tracheal occlusion reduces pulmonary hypertension in severe congenital diaphragmatic hernia. Ultrasound Obstet Gynecol. 2019 Dec;54(6):752-758. doi: 10.1002/uog.20216. Epub 2019 Nov 4. PMID 30640410
- [Background] Russo FM, Cordier AG, Basurto D, Salazar L, Litwinska E, Gomez O, Debeer A, Nevoux J, Patel S, Lewi L, Pertierra A, Aertsen M, Gratacos E, Nicolaides KH, Benachi A, Deprest J. Fetal endoscopic tracheal occlusion reverses the natural history of right-sided congenital diaphragmatic hernia: European multicenter experience. Ultrasound Obstet Gynecol. 2021 Mar;57(3):378-385. doi: 10.1002/uog.23115. PMID 32924187
- [Background] Deprest JA, Nicolaides KH, Benachi A, Gratacos E, Ryan G, Persico N, Sago H, Johnson A, Wielgos M, Berg C, Van Calster B, Russo FM; TOTAL Trial for Severe Hypoplasia Investigators. Randomized Trial of Fetal Surgery for Severe Left Diaphragmatic Hernia. N Engl J Med. 2021 Jul 8;385(2):107-118. doi: 10.1056/NEJMoa2027030. Epub 2021 Jun 8. PMID 34106556
- [Background] Deprest J, Brady P, Nicolaides K, Benachi A, Berg C, Vermeesch J, Gardener G, Gratacos E. Prenatal management of the fetus with isolated congenital diaphragmatic hernia in the era of the TOTAL trial. Semin Fetal Neonatal Med. 2014 Dec;19(6):338-48. doi: 10.1016/j.siny.2014.09.006. Epub 2014 Nov 11. PMID 25447987
- See also: CHOP Center for Fetal Diagnosis and Treatment — https://www.chop.edu/centers-programs/center-fetal-diagnosis-and-treatment
- See also: CHOP Pulmonary Hypoplasia Program — https://www.chop.edu/centers-programs/pulmonary-hypoplasia-program